CLINICAL TRIAL: NCT01607008
Title: Multiparametric MRI for Assessing Radiotherapy Treatment Response of Prostate Cancer
Brief Title: MRI for Assessing Prostate Cancer Response
Acronym: NA_00067284
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J11143; NA_00067284 (Other: JHM IRB)
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI imaging (Other): Use of MRI imaging in conjunction with standard radiation treatment
  Interventions: Other: MRI imaging

INTERVENTIONS:
Other: MRI imaging — 3 total MRI imaging studies:
  1. pre standard radiation treatment
  2. during standard radiation treatment
  3. post standard radiation treatment

SUMMARY:
Prostate cancer is one of most common cancers in America, affecting 1 in 6 men. External beam radiation therapy is one of the common methods to treat prostate cancer. Although radiotherapy is effective, side effects to the adjacent normal organs limit the therapeutic ratio. Those side effects are usually associated with the radiation damage of the normal tissue surrounding prostate, e.g. bladder, urethra and rectum etc. Both effectiveness and the side effects of radiation treatment are often accessed after whole course of radiotherapy, which makes the early intervention difficult. The current research project is a feasibility study of utilizing advanced magnetic resonance imaging (MRI) techniques to access radiotherapy treatment response of prostate cancer during and right after radiotherapy.

Many advanced MRI techniques, e.g. spectroscopy (MRS), diffusion-weighted (DWI), dynamic contrast enhanced (DCE) perfusion weighted images, have been used in radiology departments for diagnostic purpose. This research project is to study the feasibility of using advanced MRI sequences to monitor tissue response during and after radiotherapy. The tissue changes revealed from MRI can provide physicians early information on possible tumor recurrence and normal tissue toxicity, therefore, the early intervention may be possible to spare normal tissue and cure the patient. The project is designed to combine several different advanced MRI imaging techniques systematically to study tissue changes during radiotherapy, which has not been seen elsewhere to date.

Another important goal of this research project is to study the feasibility of associating functional MRI with radiation treatment dose distribution. Tissue response during radiation treatment depends on dose. The functional MRI can provide more information than simple anatomic information. Mapping the functional MRI spatially and associating them with 3D dose distribution in radiation treatment planning system is one important step to quantitative assess the relationship between radiation treatment and tissue changes due to the radiation.

DETAILED DESCRIPTION:
Twenty patients who are diagnosed with prostate cancer and will undergo external beam radiotherapy will be recruited in this study. Three MR scans of each patient under the study will be performed at different time points. Each MR scan will include several advanced MR imaging sequences (including but not limited to MR spectroscopy, diffusion and perfusion imaging, which are used in routine clinical radiology settings) in addition to typical T1 and T2 weighted MR imaging. The MR scans will be conducted at Radiation Oncology department with the position similar to the treatment position.

The first MR scan will happen prior to the radiation treatment during the scheduled patient simulation for baseline information. The T1- and T2-weighted MRI will be used for delineation of prostate gland as a part of routine treatment planning process. Additional functional MR (DWI/ADC. DCE, etc) images will be used as baseline of this study. The second MR scan with the same sequences will happen in the mid course of radiation treatment. And the third MR scan with the same sequences will happen at end of radiation treatment. Because the participated patients will come to radiation oncology department daily for their routine radiation treatment there will be no additional visits required for patients. The first scan will happen during the same day when patients undergo CT and MRI simulation for treatment planning as part of their standard cares. Two extra MRI scans will be performed as part of this research protocol. The second and third scans will happen on one of treatment days.

While it is anticipated that the advanced MRI techniques will eventually play an important role in the early intervention of radiation treatment and patient management of radiotherapy of prostate cancer at JHH, no modification of the radiation treatment and patient management will be based on the imaging information acquired during this feasibility study. All participated patients will undergo the routine radiation treatment as all other prostate cancer patients managed in our department.

The imaging data acquired will be systematically processed and analyzed along with correlating to radiation treatment dose distribution. All MRI data from three different scans need to be registered to each other and then register to planning CT. The anatomical, functional changes of tumor and normal tissues during radiation treatment will be accessed and correlated to radiation dose. After radiotherapy, all enrolled patients will be followed up the same way as normal post treatment management. The short term or long term tumor response and normal tissue side effects will also be collected under routine clinical follow up.

Following MRI based biomarker will be assessed:

* ADC map
* Dynamic contrast imaging (DCE)
* Spectroscopy
* Other MRI modalities as they are developed For example, tumor size measurement, MRI parameters of choline peak in spectroscopy, ADC values, and DCE map, tumor and normal tissue doses will be recorded for each scans. A multi-parametric analysis will be performed to seek correlations.

A new software package will be developed to help overlay the functional MRI data on top of 3D radiation dose distribution. The region of interests and the correlations between MRI data and dose will be easier to identified using under the new software. Further detail quantitative analysis can then be focused on those identified regions of interest.

Data Analysis Steps:

1. After first scan, dynamic contrast enhanced (DCE) MRI data will be processed by iCAD package to get pharmacokinetic parameters e.g. Ktrans and Ve.. A Ktrans vs Ve map will be generated. All MRI data including T1, T2, ADC map, DEC map, spectroscopy will be resampled to same resolution and registered to each other. The treatment target, prostate in this case, along with surrounding normal organs (rectum, urethral and bladder) will be delineated based on anatomical MRI images. Within prostate gland, different part of regions, cancerous or healthy regions based on functional MRI will be defined too.
2. Second and third sets of MRI scan data will be processed the same way as the Step 1 and registered to baseline scan. Same anatomical structures and same regions within prostate will be defined.
3. To test Hypothesis one, the MRI signal from the second and third scan will be compared to the baseline scan on each individual MRI sequence data and on combined all data in a multiparametric approach.The signal changes within different organs and different regions of prostate will be analyzed. A statistical significant (p<0.05) signal intensity changes within certain regions of interest can be defined as observation of signal changes.

   After kinetic and other MRI data analysis are done independently without the knowledge of the radiation dose, all registered MRI data will be imported into radiation treatment planning system. Some special software will be developed to change the some MRI data format to a recognized format for planning system. Within the treatment planning system, the MRI data will be co-registered to planning CT. The 3D dose distribution can then overlap on MRI data. The dosimetric information like maximum dose, mean dose of each organ or region of interest defined in previous steps will be calculated. The dose parameters will be calculated from stationary planning CT. There is potential dose uncertainty due to motion of prostate and rectum. However, given that external beam radiotherapy of prostate usually lasts 6-8 weeks with many fractionated treatments and image guided patient treatment ability in our clinic, the systematic organ motion is very small. Besides, most of the literature data on dose dependent tumor control and toxicity were derived from planning CT without considering organ motion. Therefore, we will not consider the effect of organ motion and use the dose parameters from stationary planning CT in this protocol.
4. The correlation between the dosimetric parameters and the signal changes will be analyzed to test the Hypothesis two.
5. Routine follow up data on tumor response (e.g PSA value) and normal tissue toxicity assessment will be collected. Although with the limited sample size of this pilot study, the direct link between MRI signal changes and treatment outcome may not be obtained. Any information, trend gathered from the correlation can be used to design next phase study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed prostate cancer
* Plan to undergo external radiation treatment of prostate cancer

Exclusion Criteria:

* Patients who cannot undergo an MRIs
* Patients who are allergic to gadolinium based contrast agent
* Patients who have cardiac pacemaker or other electronic or metal implant
* Patients who have chronic kidney disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-11-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
MRI use to predict treatment response | 2 months
  To study the feasibility of using magnetic resonance imaging (MRI) to predict treatment response in patients with prostate cancer undergoing radiation therapy. The anatomical, functional, and location changes in tumor or normal tissues during the radiation will be assessed and correlated with MRI data and treatment dose.
  Hypothesis one: Functional or anatomical MRI signal changes during the radiotherapy can be used as predictors to assess treatment response. We anticipate observing dose dependent MRI signal changes during the radiation treatment.

SECONDARY OUTCOMES:
Evaluating MRI use to predict functional radiation treatment dose distribution | 2 months
  Secondary objective: A secondary objective is evaluating the feasibility of associating functional MRI images with radiation treatment dose distribution. Both tumor control probability and normal tissue complication probability are related to the dose received by patient during the radiotherapy.
  Hypothesis two: With carefull data processing, resampling and registration, the functional MRI data can be imported into radiation treatment planning system. Quantitative analysis to assess tissue changes during radiotherapy and its correlation with radiation dose treatment can be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Danny Song, M.D., Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- The Sidney Kimmel Comprehsensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States